CLINICAL TRIAL: NCT02199236
Title: A Phase I, Dose Escalation Trial of Endoluminal High Dose Rate Brachytherapy With Concurrent Chemotherapy for Rectal or Anal Cancer in Patients With Recurrent Disease or Undergoing Non-Operative Management
Brief Title: Dose Escalation Trial of Endoluminal High-Dose-Rate Brachytherapy With Concurrent Chemotherapy for Rectal or Anal Cancer in Patients With Recurrent Disease or Undergoing Non-Operative Management
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-104
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Rectal or Anal Cancer
Keywords: High-Dose-Rate Brachytherapy; oral capecitabine; infusional 5-FU; Questionnaires; 14-104
MeSH Terms: conditions — Anus Neoplasms | interventions — Fluorouracil; Surveys and Questionnaires

ARMS (1):
- endorectal brachytherapy, concurrent chemo and questionnaires (Experimental): This is a phase I, dose-escalation study to evaluate the safety of endorectal brachytherapy with concurrent capecitabine or 5-fluoruracil (5-FU) in the management of locally recurrent/residual rectal or anal cancer in patients who have received pelvic external beam radiation therapy (EBRT) +/- chemotherapy. We will use magnetic resonance imaging (MRI) with dynamic contrast enhancement (DCE) and diffusion weighted imaging (DWI) series to contribute to the assessment of tumor response.
  Interventions: Radiation: endorectal brachytherapy; Drug: concurrent capecitabine or 5-FU; Behavioral: Questionnaires

INTERVENTIONS:
Radiation: endorectal brachytherapy — Patients will receive 3 fractions of endorectal brachytherapy, each spaced apart by 7 days (+/- 1 day). The three dose tiers will be 1500cGy (500cGy per fraction), 1800cGy (600cGy per fraction), and 2100cGy (700cGy per fraction).
Drug: concurrent capecitabine or 5-FU — Patients will receive 500 mg and 150 mg oral tablets of capecitabine for the prescribed dose of 825 mg/m2 BID, morning and evening (total daily dose of 1650 mg/m2 ). Dosages will be rounded to the nearest 150 mg or 500 mg. Tablets should be swallowed with water within 30 minutes after a meal. Capecitabine will be started on the Monday of the first week of brachytherapy (day 1) and taken on weekdays (Monday through Friday) during weeks of brachytherapy only.
  Administration of 5-FU should be only by the intravenous route taking care to avoid extravasation. Patients will receive 225 mg/m2/day, as a continuous venous infusion by a portable pump for the 3 weeks of treatment. The infusional 5-FU will be exchanged every 7 days.
Behavioral: Questionnaires — Patients should complete the 2 quality of life questionnaires during their follow-up appointments. If they are unable to be seen in follow-up, they may complete the questionnaires at home and email or mail them back to the investigator. Should there be any incomplete or ambiguous answers, a follow-up phone call will be made by a member of the research team for clarification. Additionally, if the questionnaires have not been returned within 3 weeks after the time when they are due, a member of the research team will call the patient, and the questions will be completed over the phone.
  Other Names: Bowel Function Assessment; Quality of Life Assessment

SUMMARY:
The purpose of this study is to see what amount of radiation is safe to give to rectal or anal cancer patients who are being treated with a procedure called brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally residual or recurrent cancer of the rectum or anus
* Prior pelvic EBRT
* Age > or = to 18 years
* ECOG performance status 0, 1, or 2
* At least 4 weeks from prior major surgery or radiotherapy
* Have undergone Surgical, Medical and Radiation Oncology evaluations to confirm :

  * Eligible for infusional 5-FU or capecitabine
  * Will not undergo surgery for the study disease
  * Able to receive HDR brachytherapy ANC ≥ 1.5 cells/mm3 and PLT ≥100,000/mm3
* Adequate Renal function: Creatinine <1.5 x the upper limit of normal (ULN) or calculated creatinine clearance of ≥ 50cc/min
* Adequate Hepatic functions: Bilirubin less than 1.5 mg/dL; (except in patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* AST or ALT <3xULN, or <5x ULN if known liver metastases
* Normal Cardiac function:

  * No active coronary artery disease;
  * No New York Heart Association class II, III or IV disease;
  * No arrhythmia requiring treatment
  * Maximum tumor length of 7 cm at time of brachytherapy treatment start

Exclusion Criteria:

* Women who are pregnant.
* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire treatment period and after receipt of brachytherapy. Male subjects must also agree to use effective contraception during the treatment period and until 1 year after the completion of brachytherapy.
* Patients with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study.
* Patients on concurrent anti-cancer therapy other than that allowed in the study.
* Contraindications to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 1 year
  will employ a standard 3+3 dose-escalation scheme. Patients will be accrued to the study in cohorts of 3. An initial cohort of 3 patients will be treated to each dose. The dose level will be escalated if none of the 3 patients exhibits any DLT within 90 days of completion of brachytherapy. Dose escalation will not take place until every patient in the prior dose cohort has been monitored for 90 days.

SECONDARY OUTCOMES:
tumor response | 3, 6, and 12 months
  MRI with DCE & DWI (unless contraindicated) after brachytherapy

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Wu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Follow Up Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Follow Up Only), Middletown, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow up), Commack, New York
  - Memorial Sloan Kettering Westchester (Follow Up Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Center (Follow Up Only), Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Follow-Up only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/